CLINICAL TRIAL: NCT01895621
Title: The Association of Alpha Lipoic Acid to the Median Nerve Decompression in the Carpal Tunnel Syndrome: a Randomized Controlled Trial.
Brief Title: Postoperative Alpha Lipoic Acid in the Carpal Tunnel Syndrome: a Randomized Controlled Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUNNEL ALFALIPO
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-01

CONDITIONS: Entrapment Neuropathy, Carpal Tunnel; Compression Neuropathy, Carpal Tunnel; Median Neuropathy, Carpal Tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipoic (Experimental): Median nerve decompression at the wrist, followed by Alpha lipoic acid post median nerve decompression: lipoic acid, 800 mg daily for 40 days from the day of the operation, tablets.
  Interventions: Procedure: Median nerve decompression at the wrist; Dietary Supplement: Alpha lipoic acid post median nerve decompression
- placebo (Placebo Comparator): Median nerve decompression at the wrist, followed by placebo in the same form frequency and duration as alpha lipoic acid
  Interventions: Procedure: Median nerve decompression at the wrist

INTERVENTIONS:
Procedure: Median nerve decompression at the wrist — Surgical incision of the carpal ligament at the wrist and proximal hand to decompress the median nerve.
Dietary Supplement: Alpha lipoic acid post median nerve decompression — Daily supplementation of alpha lipoic acid
  Arms: Lipoic

SUMMARY:
The postoperative course of the decompression of the median nerve in the carpal tunnel syndrome can sometimes be complicated by pain, paresthesias and other unpleasant symptoms, or may be characterized by a slow recovery of nerve function. Lipoic acid is considered to be a powerful and effective antioxidant with neuroprotective and neurotrophic properties. Dietary supplementation with lipoic acid helps reduce the damage to the nervous structure. Its action as a dietary supplement may positively modulate and accelerate healing after decompression of the median nerve.

The aim of the study is to explore any possible effects of this molecule in the postoperative period after decompression of the median nerve at the wrist.

Patients will be enrolled with proven carpal tunnel syndrome. By means of randomization, patients will be placed into one of two groups:

Group A: surgical decompression of the median nerve followed by alpha lipoic acid, 800 mg daily for 40 days.

Group B: surgical decompression of the median nerve followed by treatment with placebo

The primary endpoint of the study will be Nerve conduction velocity at 3 months after surgery after 50 days of discontinuing treatment with alpha lipoic acid (TIOBEC) / PLACEBO.

DETAILED DESCRIPTION:
The postoperative course of the decompression of the median nerve in the carpal tunnel syndrome can sometimes be complicated by pain, paresthesias and other unpleasant symptoms, or may be characterized by a slow recovery of nerve function, often also because of a prolonged illness prior to the decompression, causing extensive damage to the nerve, including demyelination, or other morphofunctional deficits. For this reason it could be particularly useful to associate a dietary supplement as a support to the structure and physiology of nerve in the post-decompression period. In this respect, the alpha-lipoic acid molecule seems to be a particularly interesting. Lipoic acid is considered to be a powerful and effective antioxidant with neuroprotective and neurotrophic properties. Dietary supplementation with lipoic acid helps reduce the damage to the nervous structure. Its action as a dietary supplement may positively modulate and accelerate healing after decompression of the median nerve.

The aim of the study is to explore any possible effects of this molecule in the postoperative period after decompression of the median nerve at the wrist.

Patients will be enrolled with proven carpal tunnel syndrome, confirmed by a careful examination including the diagnostic maneuvers Phalen, Tinel and antiPhalen. By means of randomization, patients will be placed into one of two groups:

Group A: surgical decompression of the median nerve followed by alpha lipoic acid, 800 mg daily for 40 days.

Group B: surgical decompression of the median nerve followed by treatment with placebo Surgical treatment is performed in both groups according to the standard for this type of intervention, and within 90 days after joining the waiting list.

Patients will be excluded in case of recurrent carpal tunnel syndrome. Other causes of exclusion will be carpal tunnel syndrome associated with diabetes mellitus or rheumatoid hand or secondary to other causes, uncooperative patients with poor compliance with treatment, patients with hypersensitivity to the product or one of its components, patients with pace-maker as this does not allow nerve conduction studies and electromyography, needed to evaluate pre and post treatment.

The primary endpoint of the study will be Nerve conduction velocity at 3 months after surgery after 50 days of discontinuing treatment with alpha lipoic acid (TIOBEC) / PLACEBO.

Secondary endpoints:

1. assessment of pain reported by the patient using the VAS (Visual Analogue Scale).
2. Clinical evaluation objective (presence of paresthesia and two-point discrimination on the tip of the index finger, and subjective (symptom description by the patient by means of tests and Levine-Katz questionnaire) at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

• Patients suffering from primary carpal tunnel syndrome, confirmed clinically and with nerve conduction studies

Exclusion Criteria:

* Recurrent or secondary carpal tunnel syndromes.
* Diabetic patients.
* Patients with pace-makers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Median nerve conduction velocity | Preoperatively and 90 days after median nerve decompression

SECONDARY OUTCOMES:
Score with Boston questionnaire on carpal tunnel syndrome | Preoperatively and 90 days postdecompression
Two point discrimination test on index finger pulp | Preoperatively and 90 days postdecompression

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Boriani, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy